CLINICAL TRIAL: NCT04106375
Title: Brain Mechanisms of Mindfulness Based Cognitive Therapy in Women at High Risk for Depressive Relapse ("The Women's Wellness Study")
Brief Title: Neural Effects of Wellness Classes in Women With Vulnerability to Depression ("The Women's Wellness Study")
Acronym: WWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Brain & Behavior Research Foundation (Other); Mind and Life Institute, Hadley, Massachusetts (Other); University of Arizona (Other); University of Toronto (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Marina Lopez Sola, PI of study (previously employed by CU), University of Colorado, Boulder
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-0257
Record Dates: First submitted 2019-07-09; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Major Depression
Keywords: major depression; Mindfulness based cognitive therapy; MBCT; fMRI; recurrent depression; brain
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: One group of 25 currently remitted recurrent major depression patients undergoing mindfulness based cognitive therapy for 8 weeks and one group of 25 matched healthy controls to control for time-repetition effects on brain activity and task performance
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Women with a history of depression and no other mental health disorders undergoing Mindfulness Based Cognitive Therapy.
  Interventions: Behavioral: Online mindfulness based cognitive therapy intervention
- Control (No Intervention): Healthy women with no prior history of depression or other mental health disorders as a control group for time-repetition effects on brain activity and task performance

INTERVENTIONS:
Behavioral: Online mindfulness based cognitive therapy intervention — MBCT is based on Mindfulness-Based Stress Reduction (MBSR), combining principles of cognitive therapy (CT) with those of mindfulness meditation to prevent depression relapse. Both MBSR and MBCT use contemplative practices, including sitting meditation, body scan and walking meditation, as core methods to teach awareness of negative thoughts and emotions with the aim of disengaging from pervasive patterns of ruminative self-centered mentation. Participants will be given an initial orientation session and then complete an online 8-week MBCT program. Each week participants will take part in one 2-hour online group session and will complete homework assignments anticipated to take 15-30 minutes per day to complete. Additionally, weekly phone coaching will be offered based on the modified tele-coach manual developed by Mohr and colleagues (Duffecy et al. 2010).
  Other Names: online MBCT; Mindful mood balance (MMB)
  Arms: Intervention Group

SUMMARY:
The primary objective of the study is to examine the efficacy of mindfulness based cognitive therapy (MBCT) on the prevention of relapse in women with a history of depression. Additionally, the investigators will explore how brain activity might be affected in several brain regions as a result of MBCT. This study consists of two groups, a patient group consisting of women with a history of depression and a control group consisting of healthy women. All participants within the patient group will receive an 8-week MBCT intervention program and will continue their normal medication treatment. Participants will undergo, both pre and post intervention, various behavioral and neuroimaging tasks to assess intervention effects of well-established psychological measurements related to cognitive and emotional function.

DETAILED DESCRIPTION:
Overall, this study aims to characterize the neural and psychological effects of an eight-week mindfulness based cognitive therapy (MBCT) intervention (online group class) in preventing depressive relapse in women with past history of major depression when exposed to different forms of self-relevant and context-specific emotional challenge. The investigators also aim to establish psychological and neural mechanisms contributing to depressive symptoms prior to intervention. A key objective of the study is to assess baseline markers of depressive symptoms and possible change resulting from the MBCT intervention from interdisciplinary perspectives, including the psychological perspective (i.e. measured with computer-based tasks, self-report ratings, questionnaires, etc.) and the neural perspective (neural activity measured with functional MRI).

In addition, a critical factor the investigators will be observing is the shift from more 'narrative' to 'experiential' forms of self-related awareness as a function of MBCT. Narrative self-focus refers to a concept of self that is extended in time, including past memories and intentions for the future, together with abstract self-representations in relation to socio-emotional values. In contrast, the "experiential self-focus" refers to a more immediate self-experience and is associated with greater awareness of external stimuli and internal somatic-visceral bodily states. MBSR has been shown to increase brain activity in regions relevant for conferring "experiential" self-focus (insula-opercula, dorsal anterior cingulate/supplementary motor area), while decreasing responses in rostral-medial, lateral frontal and hippocampal regions that support the "narrative" mode of self-focus. Such changes in brain activity are associated with increased well-being. Brain regions to be examined include: 1) insula-opercula and dorsal anterior cingulate brain regions responsible for mediating 'narrative' self-focus thinking styles; 2) rostral-medial and lateral frontal, and hippocampal brain regions responsible for mediating 'experiential' self-focus thinking styles; and 3) default mode and insular-paralimbic networks thought to be involved in the generation and maintenance of depressive episodes.

Behavioral Tasks

1. Breath Count Task - an objective behavioral measure of mindfulness; Dot-Probe Task - a measure of negative emotion attentional bias
2. Autobiographical Memory Interview - a means to quantify the nature of participants' autobiographical memory recall in an ecologically-valid manner
3. Free-Association Semantic Task - a measure of associative processing
4. Emotional Movies - a measure of emotional reactivity
5. N-Back Task - a measure of working memory.

Neuroimaging Tasks

1. Rest Task - a means to examine brain activity and thought content during an unconstrained task
2. 'Narrative' vs 'Experiential' Task during Autobiographical Memory Recall vs. n-back - a means to examine brain activity during 'narrative' vs 'experiential' forms of self-focus during autobiographical memory recall, vs. a demanding working memory task.
3. Self-Syllable Judgment Task - a means to examine brain activity during self-judgment vs non-self-judgment tasks.

Thought Sampling Participants will undergo an experience sampling paradigm in which daily thought surveys will be administered multiple times per day over the course of 7-10 days. These thought sampling surveys are designed to estimate several factors characterizing the occurrence of spontaneous thoughts in real-world settings as well as the nature and content of individuals' thoughts in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Women with past history of recurrent major depressive disorder

   1. Women who are not currently pregnant
   2. Meeting criteria for prior depression (at least two episodes) and showing residual symptoms of depression (PHQ-9 score of 5-12)
   3. Not meeting criteria for a current active depressive episode (SCID criteria)
   4. Having access to internet and a smartphone with data plan
   5. Receiving no antidepressant/anxiolytic medication or under a stable regime of antidepressants/anxiolytics
2. Healthy control women

   1. Women that are not currently pregnant
   2. Do not meet criteria for prior or current depression
   3. Have access to internet and a smartphone with data plan

Exclusion Criteria:

Exclusion criteria for all participants include:

* Current diagnoses of: psychosis, bipolar disorder/maniac episodes, OCD, persistent antisocial behavior, severe developmental delay, or persistent self-injury needing clinical management or therapy, organic brain injury, substance misuse.
* Past diagnoses of psychosis, bipolar disorder/mania episodes or OCD.
* Use of marijuana equal or more than 4 days per week.

Additional exclusion criteria related to Magnetic Resonance Imaging safety requirements:

We will exclude participants who have metal or electrical equipment including:

* Non-removable metal piercing
* Tattoos on head or neck, an older tattoo with metal-containing inks, and/or permanent makeup (eyeliner).
* An implanted (internal) defibrillator or pacemaker
* Cochlear (ear) implant
* Some type of clips used on brain aneurysms
* An intrauterine device (IUD) that is not compatible with the MRI scanner
* An implanted infusion pump device like an insulin pump
* Implanted nerve stimulators
* Magnetic dental appliances or fillings
* Metal plates, screws, staples, joint replacement, and prosthetics.

Additional exclusion criteria for all participants include the following:

* Clear claustrophobic symptoms.
* Abnormal capability of performing the experimental tasks as they are designed and implemented (e.g., unable to read, unable to cooperate during fMRI examination, showing visual processing impairments that cannot be corrected using lenses or any significant impairments in the processing of auditory stimulation).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Occurrence of mood episodes and post treatment relapse rate | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed via clinical interview
Depression symptoms | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed via Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001)
Rumination | Throughout study (pre-intervention to 6 months post-intervention)
  Rumination score measured using the Ruminative Response Scale (RRS; Nolen-Hoeksema 1987;1999).
Cognitive Decentering | Throughout study (pre-intervention to 6 months post-intervention)
  Score in the Experiences Questionnaire (Fresco, Moore, Dulmen, Segal, Ma, Teasdale, & Williams, 2007)
Self-Compassion | Throughout study (pre-intervention to 6 months post-intervention)
  Self-compassion scores measured using the Self-Compassion Scale (SCS: Neff, 2003).
Mindfulness | Throughout study (pre-intervention to 6 months post-intervention)
  Score on the Five-factor Mindfulness Scale (FFMQ; Baer, Smith, Hopkins, Krietemeyer & Toney, 2006)
Autobiographical Memory | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed via the Autobiographical Memory Test (Williams & Broadbent, 1986)
Self concept | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed via the Twenty Statements Test (Kuhn and McPartland, 1954)
Brain activity during autobiographical memory recall | Up to 15 weeks
  Measured using task-based fMRI bold sequence
Brain activity in the absence of a task | Up to 15 weeks
  Measured using fMRI resting-state bold sequence
Brain activity during processing of self-referential traits | Up to 15 weeks
  Measured using task-based fMRI bold sequence
Everyday thinking patterns | Up to 15 weeks
  Measured with experience sampling in daily life, questions developed for our study

SECONDARY OUTCOMES:
Mindfulness | Up to 15 weeks
  Assessed using the previously validated breath counting task (Levinson et al., 2014)
Lexical Associations | Up to 15 weeks
  Assessed using the Thought fluency task (Andrews-Hanna et al., in prep.)
Worry | Throughout study (pre-intervention to 6 months post-intervention)
  Worry score using the Penn State Worry Questionnaire (PSWQ; Meyer, Miller, Metzger, & Borkovec, 1990).
Fatigue | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed using the Multidimensional Fatigue Inventory (Smets et al. 1995).
Physical pain | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed using the Brief Pain Inventory-short form (Cleeland and Ryan, 1994).
Expectations about treatment outcome | Pre-intervention
  Score in the Credibility/Expectancy Questionnaire (CEQ, Devilly, G. J., & Borkovec, T. D. 2000)
Client satisfaction about treatment outcome | Up to 15 weeks
  Assessed using the Client Satisfaction Questionnaire (CSQ, Attkisson & Greenfield, 2009).
Positive and negative emotion | Up to 15 weeks
  Assessed by measuring responses while watching emotional movies (based on Gruber et al, 2008)
Positive and negative affect | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed using the Positive and Negative Affect Scale (PANAS; Watson & Clark, 1994)
Emotion-induced attentional bias | Up to 15 weeks
  Assessed using the dot-brobe task (Kruijt et al., 2016)
Mind wandering | Throughout study (pre-intervention to 6 months post-intervention)
  Score on the Imaginal Process Inventory (IPI, Singer et al., 1963)
Well-being | Throughout study (pre-intervention to 6 months post-intervention)
  Assessed via the Ryff Scales of Psychological Well-Being (RYFF; Ryff, 1989; Ryff & Keyes, 1995)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT04106375/Prot_000.pdf